CLINICAL TRIAL: NCT01893138
Title: A Double-blind, Randomized, Controlled Trial Comparing the Safety and Efficacy of AMDC-USR With Placebo in Female Subjects With Stress Urinary Incontinence
Brief Title: Autologous Muscle Derived Cells for Female Urinary Sphincter Repair
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cook MyoSite (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 13-003
Record Dates: First submitted 2013-07-02; First posted 2013-07-08 (Estimated); Results first posted 2023-01-05 (Actual); Last update posted 2023-01-05 (Actual); Status verified 2022-12

CONDITIONS: Stress Urinary Incontinence
Keywords: Urinary Incontinence, Stress; Tissue Therapy (Cell Therapy); Transplantation, Autologous
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo control is the vehicle solution used for the study product.
  Interventions: Other: Placebo
- Iltamiocel (Experimental): AMDC is the study product (autologous muscle-derived cells). The generic name is iltamiocel. Single intraurethral injection of 150 x 10^6 cells.
  Interventions: Biological: Iltamiocel

INTERVENTIONS:
Other: Placebo — Placebo control is the vehicle solution used for the study product.
  Arms: Placebo
Biological: Iltamiocel — AMDC is the study product (autologous muscle-derived cells). The generic name is iltamiocel. Single intraurethral injection of 150 x 10^6 cells.
  Other Names: Autologous muscle-derived cells (AMDC)
  Arms: Iltamiocel

SUMMARY:
This randomized, double-blind, placebo-controlled, multicenter, confirmatory study will evaluate the efficacy and safety of Cook MyoSite Incorporated Autologous Muscle-Derived Cells (generic name Iltamiocel) compared to a placebo (vehicle) control dose in the treatment of stress urinary incontinence (SUI) in adult female patients.

DETAILED DESCRIPTION:
Study comparing intrasphincteric injection of iltamiocel with placebo. Subjects unblinded after 12 month visits, but followed for up to 2 years. Subjects randomized to placebo could elect to receive open-label iltamiocel after completing 12 month visit.

ELIGIBILITY:
Inclusion Criteria:

* Female patient has primary symptoms of SUI, as confirmed by patient medical history and clinical symptoms, including a focused incontinence evaluation.

Exclusion Criteria:

* Patient has symptoms of pure urge incontinence as confirmed by basic evaluation of etiology from a patient medical history, including a focused incontinence history.
* Patient has symptoms of mixed urinary incontinence where urge incontinence is the predominant factor.
* Patient has had stress urinary incontinence symptoms less than 6 months prior to signing the informed consent.
* Patient has not previously attempted conservative treatment prior to signing the informed consent. (Examples of conservative treatment include behavior modifications, bladder exercises, biofeedback, etc.)
* Patient has more than 2 episode of awakening to void during normal sleeping hours.
* Patient cannot be maintained on a stable dose and/or frequency of medication (including diuretics) known to affect lower urinary tract function, including but not limited to, anticholinergics, tricyclic antidepressants or alpha-adrenergic blockers, for at least 2 weeks prior to screening or is likely to change during the course of the study.
* Patient is pregnant, lactating, or plans to become pregnant during the course of the study.
* Patient refuses to provide written informed consent.
* Patient is not at least 18 years of age.
* Patient is not available for the follow-up evaluations as required by the protocol.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 311 (Actual)
Dates: Start 2013-11-21 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2020-11-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Kaufman, M.D., Ph.D., Principal Investigator — Vanderbilt University Medical Center, Department of Urologic Surgery
Locations (29):
- United States (26):
  - Mayo Clinic Arizona Phoenix Campus, Phoenix, Arizona
  - The American Association of Female Pelvic Medicine Specialists, Agoura Hills, California
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - Stanford University, Stanford, California
  - Cleveland Clinic Florida, Weston, Florida
  - Emory University, Atlanta, Georgia
  - NorthShore University HealthSystem, Skokie, Illinois
  - IU Health Physicians Urogynecology, Indianapolis, Indiana
  - Female Pelvic Medicine & Urogynecology Institute of Michigan, Grand Rapids, Michigan
  - Mercy Health Saint Mary's Campus, Grand Rapids, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - NYU Urology Associates, New York, New York
  - Premier Medical Group of the Hudson Valley PC, Poughkeepsie, New York
  - Montefiore Medical Center, The Bronx, New York
  - McKay Urology, Charlotte, North Carolina
  - The Carl and Edyth Lindner Center for Research and Education at The Christ Hospital, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Greenville Health System, Greenville, South Carolina
  - Sanford Female Pelvic Medicine and Reconstructive Surgery Clinic, Sioux Falls, South Dakota
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Methodist Urology Associates, Houston, Texas
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Benaroya Research Institute at Virginia Mason, Seattle, Washington
- University Hospital Leuven, Leuven, Belgium
- Germany (2):
  - Universitätsklinikum Essen, Essen
  - Praxisklinik Urologie Rhein-Ruhr (PUR/R), Mülheim

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kaufman MR, Goldman HB, Chermansky CJ, Dmochowski R, Kennelly MJ, Peters KM, Quiroz LH, Bennett JB, Thomas S, Marguet CG, Benson KD, Lee UJ, Sokol ER, Wolter CE, Katz DM, Tarnay CM, Antosh D, Heit MH, Rehme C, Karram M, Snyder S, Canestrari E, Jankowski RJ, Chancellor MB. Iltamiocel Autologous Cell Therapy for the Treatment of Female Stress Urinary Incontinence: A Double-Blind, Randomized, Stratified, Placebo-Controlled Trial. Neurourol Urodyn. 2024 Nov;43(8):2290-2299. doi: 10.1002/nau.25588. Epub 2024 Sep 16. PMID 39282854
- [Derived] Antosh DD, High R, Brown HW, Oliphant SS, Abed H, Philip N, Grimes CL. Feasibility of prophylactic salpingectomy during vaginal hysterectomy. Am J Obstet Gynecol. 2017 Nov;217(5):605.e1-605.e5. doi: 10.1016/j.ajog.2017.07.017. Epub 2017 Jul 20. PMID 28734829

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 311 subjects were enrolled (underwent biopsy procedure) and 297 subjects underwent study treatment with iltamiocel (199 subjects) or placebo (98 subjects). Analysis population is based on 297 subjects that underwent study treatment. At randomization, participants stratified by presence or absence of prior incontinence surgery and by < 10 or ≥10 stress incontinence episodes over 3 day diary at screening.
Groups:
- Placebo: Placebo control is the vehicle solution used for the study product. Single intraurethral injection of vehicle control.
Period: Double-Blind Period
Arm/Group | Iltamiocel | Placebo
Started | 199 | 98
Injection | 199 | 98
1 Month Follow-Up | 199 | 97
3 Month Follow-Up | 199 | 97
6 Month Follow-Up | 198 | 97
12 Month Follow-Up | 198 | 97
Completed | 198 | 97
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1
Period: Open Label - Unblinded Period
Arm/Group | Iltamiocel | Placebo
Started | 198 | 97
Open Label Period | 166 | 97
Iltamiocel Injection (No additional treatment for iltamiocel arm. Subjects originally randomized to placebo received single, open-label iltamiocel injection.) | 0 | 92
2 Year Follow-Up | 166 | 87
Completed | 166 | 87
Not Completed | 32 | 10
Not completed — Lack of Efficacy | 9 | 0
Not completed — Lost to Follow-up | 4 | 3
Not completed — Withdrawal by Subject | 18 | 7
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Population: Women ≥18 years or older with stress-predominant urinary incontinence.
Groups:
- Total: Total of all reporting groups
Arm/Group | Iltamiocel | Placebo | Total
Number analyzed (Participants) | 199 | 98 | 297
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.1 (10.9) | 55.0 (10.7) | 54.4 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 199 | 98 | 297
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 5 | 8
  Not Hispanic or Latino | 196 | 93 | 289
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 0 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 3 | 8
  White | 184 | 89 | 273
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 3 | 5 | 8
Region of Enrollment [Number; unit: participants]
  Belgium | 2 | 1 | 3
  United States | 193 | 94 | 287
  Germany | 4 | 3 | 7
Stress Incontinence Episodes Over 3 Day Diary [Mean (Standard Deviation); unit: stress leaks] — Participant recorded number of stress leaks over 3 days in electronic diary.
  stress leaks | 14.2 (9.8) | 15 (14.2) | 14.5 (11.4)
24 Hour Pad Test Weight [Mean (Standard Deviation); unit: grams] — A test in which the participant wears specific absorbent pads dispensed by the clinic. The pads are weighed to record the pre-test weight prior to dispensing to the participant. The participant must wear the absorbent pads for 24 hours. The participant returns the used absorbent pads to the clinic, and the clinic records the post-test weight to determine urinary leakage for the 24 hour period. The difference in weights represent the amount of urine leaked in which 24 hour pad weight = total weight of pads after test period - total weight of pads prior to test period.
  grams | 47.6 (91.8) | 40.9 (52.8) | 45.2 (81.1)
Incontinence Quality of Life (IQOL) Assessment -Total Score [Mean (Standard Deviation); unit: scores on scales] — The I-QOL questionnaire is a validated, 22-item tool used to assess quality of life (QOL) of women with urinary incontinence, focused on avoidance and limiting behavior, psychosocial impacts, and social embarrassment. Score scale is 0-100; increased score indicates improvement.. Scored 0 to100, with higher scores indicating a better QOL
  scores on scales | 59.0 (21.0) | 59.5 (20.2) | 59.2 (20.0)
7-Item Incontinence Impact Questionnaire - Short Form (IIQ-7) [Mean (Standard Deviation); unit: scores on scales] — The IIQ-7 questionnaire is a validated, 7-item tool used to assess the impact of urinary incontinence on health-related quality of life, focused on physical activity, social relationships, travel, and emotional health. Scored 0 to 100, lower scores indicate better quality of life (QOL).
  scores on scales | 44.4 (20.9) | 43.7 (21.8) | 44.2 (21.2)
6-Item Urogenital Distress Inventory Score - Short Form (UDI-6) [Mean (Standard Deviation); unit: scores on scales] — This questionnaire consists of 6 questions focused on symptoms related to stress urinary incontinence, detrusor overactivity, and bladder outlet obstruction. Score scale is 0-75; decreased score indicates improvement.
  scores on scales | 38.5 (16) | 40.5 (18.4) | 39.2 (16.8)
Global Quality of Life Assessment (GQOL) [Mean (Standard Deviation); unit: scores on scales] — This questionnaire consists of 1 question focused on satisfaction with condition. Score scale is 0-6; decreased score indicates improvement.
  scores on scales | 5.7 (1.0) | 5.6 (1.1) | 5.7 (1.0)
Incontinence Severity Index (ISI) [Mean (Standard Deviation); unit: scores on scales] — The ISI is a questionnaire consisting of two questions which assesses the frequency and quantity of urine leakage. Score scale is 0-12; decreased score indicates improvement.
  scores on scales | 7.6 (2.4) | 7.4 (2.8) | 7.5 (2.5)

OUTCOME MEASURES:

1. Primary Outcome: Participants With ≥ 50% Reduction in Stress Incontinence Episode Frequency From Baseline to 12 Months Post-treatment; as Assessed by 3 Day Diary
Time Frame: Baseline and 12 months
Population: All participants with baseline and 12 month 3 day diary data
Measure: Count of Participants; unit: Participants
Arm/Group | Iltamiocel | Placebo
Number analyzed (Participants) | 198 | 97
Participants | 103 | 52

2. Secondary Outcome: Participants With at ≥ 75% Reduction in Stress Incontinence Episodes From Baseline at 12 Months
Time Frame: Baseline and 12 months
Population: All participants with baseline and 12 month 3 day diary data
Measure: Count of Participants; unit: Participants
Arm/Group | Iltamiocel | Placebo
Number analyzed (Participants) | 198 | 97
Participants | 73 | 30

3. Secondary Outcome: Participants With 0 or 1 Stress Incontinence Episodes Based on 3 Day Diary Records at 12 Months
Time Frame: Baseline and 12 months
Population: All participants with baseline and 12 month diary data
Measure: Count of Participants; unit: Participants
Arm/Group | Iltamiocel | Placebo
Number analyzed (Participants) | 198 | 97
Participants | 53 | 22

4. Secondary Outcome: Change in the Frequency of Stress Incontinence Episodes From Baseline at 12 Months
Time Frame: Baseline and 12 months
Population: All participants with baseline and 12 month 3 day diary data
Measure: Mean (Standard Deviation); unit: stress leaks
Arm/Group | Iltamiocel | Placebo
Number analyzed (Participants) | 198 | 97
stress leaks | -5.8 (11) | -4.9 (13.5)

5. Other Pre Specified Outcome: Association of Change in Quality of Life Scores With Change in Stress Incontinence Episode Frequency
Description: Spearman's correlation used for analysis
Time Frame: Baseline and 12 months
Population: All participants with baseline and 12 month diary data
Measure: Number; unit: correlation coefficient
Arm/Group | Iltamiocel | Placebo
Number analyzed (Participants) | 198 | 96
correlation coefficient
  Association of IQOL improvement with stress incontinence episode reduction at 12 months | -0.556 | -0.456
  Association of IIQ-7 improvement with stress incontinence episode reduction at 12 months | 0.522 | 0.442
  Association of UDI-6 improvement with stress incontinence episode reduction at 12 months | 0.408 | 0.433
  Association of GQOL improvement with stress incontinence episode reduction at 12 months | 0.537 | 0.422
  Association of ISI improvement with stress incontinence episode reduction at 12 months | 0.529 | 0.599

6. Other Pre Specified Outcome: Treatment Durability at 24 Months
Description: Treatment durability defined as iltamiocel-treated participants with reduction in stress incontinence episode frequency (SIEF) at 12 months who maintained that response at 24 months
Time Frame: Baseline, 12 months, and 24 months after injection with iltamiocel
Population: All participants who received iltamiocel treatment during the double-blind period and with 12-month and 24-month stress incontinence episode frequency (SIEF) diary data. Participants who received placebo treatment in the double-blind period are not included due to receiving iltamiocel treatment in the open-label period after unblinding or were exited from the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Iltamiocel
Number analyzed (Participants) | 199
Participants
  Participants that had ≥ 50% reduction in stress incontinence episodes at Month 12 and Month 24 data: number analyzed (Participants) | 89
  Participants that had ≥ 50% reduction in stress incontinence episodes at Month 12 and Month 24 data | 80
  Participants that had ≥ 75% reduction in stress incontinence episodes at Month 12 and Month 24 data: number analyzed (Participants) | 65
  Participants that had ≥ 75% reduction in stress incontinence episodes at Month 12 and Month 24 data | 50
  Participants that had ≤1 stress incontinence episodes at Month 12 and Month 24 data: number analyzed (Participants) | 45
  Participants that had ≤1 stress incontinence episodes at Month 12 and Month 24 data | 36

7. Post Hoc Outcome: Participants With at ≥ 75% Reduction in Stress Incontinence Episodes From Baseline at 12 Months (Prior Surgery Participants Only)
Description: Participants with a history of prior SUI surgery with baseline and 12 month diary data.
Time Frame: Baseline and 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Iltamiocel | Placebo
Number analyzed (Participants) | 50 | 25
Participants | 20 | 4

8. Post Hoc Outcome: Participants With 0 or 1 Stress Incontinence Episodes Based on 3 Day Diary Records at 12 Months (Prior Surgery Participants Only)
Description: Participants with a history of prior SUI surgery with baseline and 12 month diary data.
Time Frame: Baseline and 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Iltamiocel | Placebo
Number analyzed (Participants) | 50 | 25
Participants | 14 | 3

9. Post Hoc Outcome: Change in the Frequency of Stress Incontinence Episodes From Baseline at 12 Months (Prior Surgery Participants Only)
Description: Participants with a history of prior SUI surgery with baseline and 12 month diary data.
Time Frame: Baseline and 12 months
Measure: Mean (Standard Deviation); unit: stress leaks
Arm/Group | Iltamiocel | Placebo
Number analyzed (Participants) | 50 | 25
stress leaks | -6.7 (14.5) | -4.5 (11.5)

10. Post Hoc Outcome: Association of Change in Quality of Life Scores With Change in Stress Incontinence Episode Frequency (Prior Surgery Participants Only)
Description: Spearman's correlation used for analysis
Time Frame: Baseline and 12 months
Population: All participants with prior surgery and baseline and 12 month diary data
Measure: Number; unit: correlation coefficient
Arm/Group | Iltamiocel | Placebo
Number analyzed (Participants) | 50 | 25
correlation coefficient
  Association of IQOL improvement with stress incontinence episode reduction at 12 months | -0.489 | -0.460
  Association of IIQ-7 improvement with stress incontinence episode reduction at 12 months | 0.427 | 0.542
  Association of UDI-6 improvement with stress incontinence episode reduction at 12 months | 0.424 | 0.604
  Association of GQOL improvement with stress incontinence episode reduction at 12 months | 0.561 | 0.190
  Association of ISI improvement with stress incontinence episode reduction at 12 months | 0.426 | 0.476

11. Post Hoc Outcome: Treatment Durability at 24 Months (Prior Surgery Participants)
Description: Treatment durability defined as participants with reduction in stress incontinence episode frequency (SIEF) at 12 months who maintained response at 24 months
Time Frame: Baseline, 12 months, and 24 months after injection with iltamiocel
Population: Prior surgery participants who received iltamiocel treatment during the double-blind period with 12-month and 24-month stress incontinence episode frequency (SIEF) diary data. Prior surgery participants who received placebo treatment in the double-blind period are not included due to receiving iltamiocel treatment in the open-label period after unblinding or were exited from the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Iltamiocel
Number analyzed (Participants) | 53
Participants
  Participants that had ≥ 50% reduction in stress incontinence episodes at Month 12 and Month 24 data: number analyzed (Participants) | 22
  Participants that had ≥ 50% reduction in stress incontinence episodes at Month 12 and Month 24 data | 19
  Participants that had ≥ 75% reduction in stress incontinence episodes at Month 12 and Month 24 data: number analyzed (Participants) | 18
  Participants that had ≥ 75% reduction in stress incontinence episodes at Month 12 and Month 24 data | 12
  Participants that had ≤1 stress incontinence episodes at Month 12 and Month 24 data: number analyzed (Participants) | 13
  Participants that had ≤1 stress incontinence episodes at Month 12 and Month 24 data | 11

ADVERSE EVENTS:
Time Frame: 12 month double-blind period and open label unblinded period from month 12 to 24
Description: Collection at biopsy, injection, 1 month, 3 months, 6 months, and 12 months post-treatment for double-blind period for comparison between treatment arms prior to unblinding investigator and participant. Subjects unblinded after 12 month visit, but followed for up to 2 years. Subjects randomized to placebo could elect to receive open-label iltamiocel after completing 12 month visit.
Groups:
- Iltamiocel - Double-Blind Period: AMDC is the study product (autologous muscle-derived cells). The generic name is iltamiocel. Single intraurethral injection of 150 x 10^6 cells.
- Placebo - Double-Blind Period: Placebo control is the vehicle solution used for the study product. Single intraurethral injection of vehicle control.
- Iltamiocel - Unblinded Period: Subjects who received iltamiocel in double-blind period. No additional treatment for iltamiocel arm in unblinded period.
- Placebo Receiving Open Label Iltamiocel in Unblinded Period: Subjects who received placebo in double-blind period and elected to receive iltamiocel injection in unblinded period. Single intraurethral injection of 150 x 10^6 cells.
Arm/Group | Iltamiocel - Double-Blind Period | Placebo - Double-Blind Period | Iltamiocel - Unblinded Period | Placebo Receiving Open Label Iltamiocel in Unblinded Period
All-Cause Mortality (participants affected / at risk) | 0/199 | 0/98 | 0/198 | 0/92
Serious Adverse Events (participants affected / at risk) | 11/199 | 9/98 | 12/198 | 4/92
Other Adverse Events (participants affected / at risk) | 84/199 | 28/98 | 21/198 | 22/92
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Iltamiocel - Double-Blind Period (N=199) | Placebo - Double-Blind Period (N=98) | Iltamiocel - Unblinded Period (N=198) | Placebo Receiving Open Label Iltamiocel in Unblinded Period (N=92)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Coronary artery dissection (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Related to Iltamiocel and Injection Procedure
Sepsis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Staphylococcal infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Scoliosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Major depression (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Procedural Pain (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0) — Related to Biopsy Procedure
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bacteremia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infectious pleural effusion (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia staphylococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intentional Overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Joint lock (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Panic attack (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malignant hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Subgaleal haematoma (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Iltamiocel - Double-Blind Period (N=199) | Placebo - Double-Blind Period (N=98) | Iltamiocel - Unblinded Period (N=198) | Placebo Receiving Open Label Iltamiocel in Unblinded Period (N=92)
Injection site pain (General disorders) | 10 (11) | 1 (1) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 36 (53) | 14 (19) | 14 (16) | 10 (12)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (8) | 5 (6) | 2 (2) | 3 (3)
Dysuria (Renal and urinary disorders) | 20 (20) | 7 (8) | 1 (1) | 6 (6)
Sinusitis (Infections and infestations) | 11 (11) | 1 (1) | 4 (4) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-02-18): https://cdn.clinicaltrials.gov/large-docs/38/NCT01893138/Prot_SAP_000.pdf